CLINICAL TRIAL: NCT04609709
Title: Thrust Manipulation, Electric Dry Needling and Exercise Vs. Non-thrust Mobilization, Soft-Tissue Mobilization, Exercise and TENS for Tension Type Headache Sufferers
Brief Title: HVLAT, Electric DN, Exercise Vs. Mobilization, STM, Exercise, TENS for Tension Type Headaches
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alabama Physical Therapy & Acupuncture (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, James Dunning, DPT, MSc, FAAOMPT, DPT, MSc, FAAOMPT, Alabama Physical Therapy & Acupuncture
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAMT51
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Tension-Type Headache
MeSH Terms: conditions — Tension-Type Headache | interventions — Exercise; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- thrust manipulation, electric dry needling and exercise (Experimental): thrust manipulation, electric dry needling and exercise
  Interventions: Other: Thrust Manipulation, Electric Dry Needling and Exercise
- non-thrust Mobilization, Soft-Tissue Mobilization, Exercise and TENS (Active Comparator): non-thrust mobilization, soft-tissue mobilization, exercise and TENS
  Interventions: Other: Non-thrust Mobilization, Soft-Tissue Mobilization, Exercise and TENS

INTERVENTIONS:
Other: Thrust Manipulation, Electric Dry Needling and Exercise — Thrust Manipulation, Electric Dry Needling
  Arms: thrust manipulation, electric dry needling and exercise
Other: Non-thrust Mobilization, Soft-Tissue Mobilization, Exercise and TENS — Non-thrust Mobilization, Soft-Tissue Mobilization, Exercise and TENS
  Arms: non-thrust Mobilization, Soft-Tissue Mobilization, Exercise and TENS

SUMMARY:
The purpose of this research is to compare two different approaches for treating patients with tension-type headaches: thrust Manipulation, electric dry Needling and exercise Vs. non-thrust mobilization, soft-tissue mobilization, exercise and TENS. Physical therapists commonly use all of these techniques to treat tension-type headaches. This study is attempting to find out if one treatment strategy is more effective than the other.

DETAILED DESCRIPTION:
Patient will tension-type headaches will be randomized to receive 2 sessions per week for 6 weeks (up to 8-12 sessions total) of either: 1. thrust Manipulation, electric dry Needling and exercise or 2. non-thrust mobilization, soft-tissue mobilization, exercise and TENS

ELIGIBILITY:
Inclusion Criteria:

* Patient must be between 18 and 65 years old and report ALL YES under one of the Tension-type Headaches described below:

2.2 Frequent Episodic Tension-type Headaches: Frequent episodes of headache, typically bilateral, pressing or tightening in quality and of mild to moderate intensity, lasting minutes to days. The pain does not worsen with routine physical activity and is not associated with nausea, but photophobia or phonophobia may be present.

1. At least 10 episodes of headache occurring on 1- 14 days per month on average for >3 months (12 and <180 days per year)
2. Headache lasting from 30 minutes to 7 days
3. Patient has headaches that have at least two of the following four characteristics:

   1. Bilateral location
   2. Pressing or tightening (non-pulsating) quality
   3. Mild or moderate intensity
   4. Not aggravated by routine physical activity such as walking or climbing stairs
4. Both of the following are true:

   1. No nausea or vomiting
   2. No more than one of photophobia or phonophobia

2.2.1 Frequent Episodic Tension-type Headache associated with pericranial tenderness

1. Episodes fulfilling criteria for Frequent episodic tension-type headache (See 2.2 above)
2. Increased pericranial tenderness on manual palpation.

2.3 Chronic Tension-type Headaches: A disorder evolving from frequent episodic tension-type headache, with daily or very frequent episodes of headache, typically bilateral, pressing or tightening in quality and of mild to moderate intensity, lasting hours to days, or unremitting. The pain does not worsen with routine physical activity, but may be associated with mild nausea, photophobia or phonophobia.

1. Headache occurring on 15 days per month on average for >3 months (180 days per year)
2. Headache lasting hours to days, or unremitting
3. At least two of the following four characteristics

   1. Bilateral location
   2. Pressing or tightening (non-pulsating) quality
   3. Mild or moderate intensity
   4. Not aggravated by routine physical activity such as walking of climbing stairs
4. Both of the following:

   1. No more than one of the photophobia, phonophonbia, or mild nausea
   2. Neither moderate or severe nausea nor vomiting

2.3.1 Chronic Tension-type Headache associated with pericranial tenderness

1. Headache fulfilling criteria for 2.3 Chronic tension- type headache
2. Increased pericranial tenderness on manual palpation.

Exclusion Criteria:

Exclusion Criteria: Must all be NO to be eligible

1. Patient presents with other primary and/or secondary headache
2. Patient presents with Medication Overuse Headache defined as:

   1. Headache occurring on 15 days per month in a patient with a pre-existing headache disorder
   2. Regular overuse for >3 months of one of more drug that can be taken for acute and/or symptomatic treatment of headache
   3. Not better accounted for by another headache diagnosis
3. History of head/neck trauma (to include whiplash)
4. History of Cervical Stenosis
5. Presence of any of the following atherosclerotic risk factors: hypertension, diabetes, heart disease, stroke, transient ischemic attack, peripheral vascular disease, smoking, hypercholesterolemia or hyperlipidemia
6. Red flags noted in the patient's Neck Medical Screening Questionnaire (i.e. tumors, fracture, metabolic diseases, RA, osteoporosis, history of prolonged steroid use, etc.
7. Bilateral upper extremity symptoms
8. Evidence of CNS involvement, to include hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes).
9. Two or more positive neurologic signs consistent with nerve root compression, including any 2 of the following:

   1. Muscle weakness involving a major muscle group of the upper extremity.
   2. Diminished UE deep tendon reflex of the biceps, brachioradialis, triceps or superficial flexors
   3. Diminished or absent sensation to pinprick in any UE dermatome.
10. Prior surgery to neck of thoracic spine
11. Involvement in litigation or worker's compensation regarding their neck pain and/or headaches
12. Diagnosis of fibromyalgia syndrome
13. Received anesthetic blocks or botulinum toxin within the previous 6 months
14. Received physical treatment in the neck and head the previous 6 months
15. Any condition that might contraindicate spinal manipulative therapy
16. Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-10-31 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Headache Intensity (NPRS) | Baseline, 4-weeks, 8-weeks, 12-weeks
  Average Numeric Pain Rating Score. Higher score means greater pain

SECONDARY OUTCOMES:
Change in Headache Disability Inventory | Baseline (4-Weeks After Initial Evaluation, but BEFORE the first treatment is given), 4-weeks, 8-weeks, 12-weeks
  25 questions each worth 0-4 points with maximum score of 100 points possible. Greater scores indicate increased disability.
Change in GROC (Global Rating of Change score) | 8 Weeks, 12 weeks
  GROC (ranges from -7 to +7). Global Rating of Change score.
Change in Headache Frequency | Baseline (4-Weeks After Initial Evaluation, but BEFORE the first treatment is given), 4-weeks, 8-weeks, 12-weeks
  Number of days patient has a headache during last time period
Change in Headache Duration | Baseline (4-Weeks After Initial Evaluation, but BEFORE the first treatment is given), 4-weeks, 8-weeks, 12-weeks
  Average number of hours/day that the patient had a headache during last time period
Change in Medication Intake (Frequency of medication intake during last time period) | Baseline, 3-months
  Frequency of medication intake during last time period

CONTACTS AND LOCATIONS:
Overall Officials: James Dunning, DPT PhD, Principal Investigator — American Academy of Manipulative Therapy
Locations (1):
- Maller and Swoverland Orthopedic PT, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided